CLINICAL TRIAL: NCT03487640
Title: Laparoscopica Hindgut Resection Plus Rectum Suspention Compare With Transanal Rectal Mucosa Resection for ODS With Rectal Prolapse
Brief Title: Surgical Treatment for ODS With Rectal Prolapse Surgical Treatment for Rectal Prolapse
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Third Military Medical University, Third Military Medical University
Other Study IDs: LarTARP
Record Dates: First submitted 2018-01-29; First posted 2018-04-04 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Constipation by Outlet Obstruction
Keywords: constipation, surgery
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transanal rectal mucosa resection: TARMR: Transanal resection of rectal mucosa for at least 5cm in length.
  Interventions: Procedure: TARMR
- Laparoscopic rectal suspension and colectomy: LARSC: We are going to suspend the rectum and to resect rigmarole hidgut Laparoscopically
  Interventions: Procedure: LARSC

INTERVENTIONS:
Procedure: TARMR — Transanal resection of rectal mucosa for at least 5cm in length.
  Groups: Transanal rectal mucosa resection
Procedure: LARSC — We are going to suspend the rectum and to resect rigmarole hidgut Laparoscopically
  Groups: Laparoscopic rectal suspension and colectomy

SUMMARY:
Chronic obstinate constipation is hard to deal with in clinic. Especially for obstructed defecation syndrome(ODS). Rectal prolapse is the most common type of ODS. Lots of surgical procedures have been suggested for it but with unsatisfactory results.To develop new surgical treatment and to provide higher quality proof for this intractable condition is of significance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ODS by defecography, coloscopy, barium enema and dynamic MRI.
* Patients should accord with Rome IV criteria.

Exclusion Criteria:

* Severe heart or other organ disease.
* test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meet for Rome IV criteria for constipation.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Wexner constipation score | 2019.1-2019.12
  The Wexner constipation score should be filled out
patients' satisfaction rate | 2019.1-2019.12
  The researcher will statistic the satisfaction rate of the patients

SECONDARY OUTCOMES:
short period complications | 2018.1-2019.12
  postoperative 30-day complications
operative time | 2018.1-2019.12
  the total operative time
quality of life | 2019.1-2019.12
  SF-36 form

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yang, Dr., Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Weidong Tong, Yuzhong, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No